CLINICAL TRIAL: NCT05169970
Title: A Phase II Study of Decipher-Guided Dose Escalated Radiation Therapy In Unfavorable Intermediate Risk Prostate Cancer Patients Treated SBRT Alone Without Androgen Deprivation Therapy
Brief Title: A Study of Stereotactic Body Radiation Therapy (SBRT) Without Androgen Deprivation Therapy (ADT) in People With Unfavorable Intermediate-Risk Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-458
Record Dates: First submitted 2021-12-09; First posted 2021-12-27 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Unfavorable Intermediate-Risk Prostate Cancer; Stereotactic Body Radiation Therapy (SBRT); 21-458
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a phase II nonrandomized noninferiority trial that aims to evaluate the efficacy of dose escalated radiation therapy in the absence of androgen deprivation therapy for Decipher genomic score stratified NCCN unfavorable intermediate risk prostate cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with low-intermediate risk Decipher scores (Experimental): Will receive ultrahypofractionated EBRT to the prostate and seminal vesicles (40Gy in 5 fractions).
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Patients with high risk Decipher scores (Experimental): Will receive ultrahypofractionated EBRT to the prostate and seminal vesicles (40Gy in 5 fractions) with a boost of up to 45Gy to the dominant intraprostatic lesion as identified on pretreatment MRI plus hypofractionated pelvic EBRT (25Gy in 5 fractions).
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients with a low or intermediate risk Decipher score will receive radiation targeting the seminal prostate and seminal vesicles to a dose of 40 Gy in 5 fractions delivered every other day.
  Arms: Patients with low-intermediate risk Decipher scores
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients with high risk Decipher scores will receive radiation targeting the prostate and seminal vesicles to a dose of 40 Gy in 5 fractions with a simultaneous integrated boost to 45 Gy of any dominant intraprostatic lesion as well as radiation to the pelvic lymph nodes to a dose of 25 Gy in 5 fractions delivered every other day.
  Arms: Patients with high risk Decipher scores

SUMMARY:
The researchers are doing this study to find out if stereotactic body radiation therapy (SBRT) without androgen deprivation therapy (ADT) is an effective treatment approach for people with unfavorable intermediate-risk prostate. The researchers will see whether SBRT can prevent participants' cancer from coming back and/or spreading to other parts of the body. In addition, they will look closely at how safe and effective it is to rely on Decipher test results for determining which patients would benefit from more extensive radiation treatments

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of prostate adenocarcinoma within 12 months of enrollment
* Unfavorable intermediate risk prostate cancer by NCCN 2021 risk stratification guidelines, including any of the following clinicopathologic features:
* Gleason Score 4+3
* ≥ 50% biopsy cores positive
* Two or more of the following risk factors:

  * Grade Group 2 or 3
  * cT2b-T2c
  * PSA 10 - 20 ng/mL
* Able to undergo MRI for initial staging and MR based radiation planning
* Sufficient biopsy tissue available for Decipher genomic testing
* Prostate volume < 90cc
* IPSS ≤ 20
* Age ≥ 18
* KPS ≥ or ECOG 0-2
* Estimated life expectancy >5 years
* Willing and able to provide written informed consent and Authorization for Use and Release of Health and Research Study Information (HIPAA authorization)

Exclusion Criteria:

* Radiographic T3-T4 detected on staging mpMRI

  °Must be "consistent with" (>90% probability) or suspicious for/probable/probably (75%-90% probability) ofT3-T4 disease determined by the reading radiologist.
* Evidence of distant metastases as determined by MRI, PET, or CT imaging
* Evidence of pelvic lymph node involvement as determined by MRI, PET, or CT imaging
* Prior treatment for prostate cancer including chemotherapy, surgery, or hormonal therapy
* Prior pelvic radiation
* Active second malignancy or past history of malignancies diagnosed within the last 2 years that requires active therapy and/or in remission, with the exception of resected non-melanoma skin cancers, non-muscle invasive bladder cancer, stage I head and neck cancer, or stage I colorectal cancer
* TURP or greenlight PVP within 6 months of enrollment
* History of Crohn's Disease or Ulcerative Colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 215 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of biochemical progression free survival | 2 years
  Biochemical progression will be determined according to the established criteria of 2 ng/nl elevation of the PSA nadir level (nadir + 2 definition).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gorovets, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm